CLINICAL TRIAL: NCT05556798
Title: Belantamab Mafodotin in Combination With Nirogacestat and Pomalidomide in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Belantamab Mafodotin in Combination With Nirogacestat and Pomalidomide in People With Multiple Myeloma That Has Not Responded to Treatment or Has Come Back After Treatment
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-495
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Belantamab Mafodotin; Nirogacestat; 21-495; Memorial Sloan Kettering Cancer Center; Pomalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; nirogacestat; pomalidomide

STUDY DESIGN:
Intervention Model Description: This is a phase Ib study with trial treatment is a combination of belantamab mafodotin (GSK2857916) and nirogacestat. A standard 3+3 dose escalation design with three planned doses of belantamab mafodotin will be implemented. There will be a 1:1 randomization between nirogacestat 100 mg BID or 100 mg QD during the 4 day run-in period prior to starting belantamab mafodotin on Cycle 1 Day 1 (days -4 to -1).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belantamab Mafodotin and Nirogacestat (Experimental): There will be a 1:1 randomization betweennirogacestat 100 mg BID or 100 mg QD during the 4day run-in period prior to starting belantamab mafodotin on Cycle 1 Day 1 (days -4 to -1). The cycle length for Cycles 1-3 is 21 days (3 weeks). Treatment with nirogacestat will be 100 mg BID continuously during each cycle for all subjects. Belantamab mafodotin will be administered via IV infusion in an outpatient setting on Day 1 of Cycles 1-3 and nirogacestat 100mg BID will be administered continuously on Days 1-21 of each cycle. Treatment with belantamab mafodotin will be given at an initial dose of 1.0 mg/kg. The study will have a 3+3 dose escalation design for belantamab mafodotin. Belantamab mafodotin dose levels are 1.0 mg/kg, 1.4 mg/kg, and 1.9 mg/kg. Pomalidomide was added, 2 mg to the 1.4 mg/kg and 1.9 mg/kg dose cohorts.
  Interventions: Drug: Belantamab Mafodotin; Drug: Nirogacestat; Drug: Pomalidomide

INTERVENTIONS:
Drug: Belantamab Mafodotin — Belantamab mafodotin will be administered via IV infusion in an outpatient setting on Day 1 of Cycles 1-3. Treatment with belantamab mafodotin will be given at an initial dose of 1.0 mg/kg. The study will have a 3+3 dose escalation design for belantamab mafodotin. Belantamab mafodotin dose levels are 1.0 mg/kg, 1.4 mg/kg, and 1.9 mg/kg
  Other Names: GSK2857916
Drug: Nirogacestat — 1:1 randomization between nirogacestat 100mg BID or 100 mg QD during the 4 day run-in period. Treatment with nirogacestat will be 100mg BID continuously during each cycle for all subjects.
Drug: Pomalidomide — After the 4-day run-in period, all patients will receive nirogacestat in combination with belantamab, mafodotin and pomalidomide. Pomalidomide was added for day 1-14 for cycle 1-3 and day 1-14 and day 21-35 for C4+.

SUMMARY:
The purpose of this study is to find out whether combination treatment with the study drugs belantamab mafodotin, nirogacestat, and pomalidomide is a safe treatment for people who have relapsed or refractory multiple myeloma. The researchers will test different doses of belantamab mafodotin to find the safest dose to give with nirogacestat and pomalidomide. The researchers also want to find out whether belantamab mafodotin plus nirogacestat and pomalidomide is an effective treatment for this type of bone marrow cancer, and the researchers will do tests that show whether the study treatment slows or stops the growth of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory multiple myeloma treated with 3 or more prior lines of therapy. Relapsed/refractory multiple myeloma is defined by the International Myeloma Working Group (IMWG) updated criteria.
* Patients need to have measurable disease defined by one or more of the following:

  1. Serum myeloma (M)-protein greater than or equal to 0.5 g/dL (5 g/L).
  2. Urine M-protein ≥ 200 mg/24 h.
  3. Involved free light chain level ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65). Measurable plasmacytoma(s) verified by imaging or biopsy (≥1 lesion that has a single diameter of ≥2cm)

  e. A bone marrow biopsy demonstrating ≥30% infiltration of clonal plasma cells verified by CD138 immunohistochemistry.
* Have undergone autologous stem cell transplant or are considered transplant ineligible.
* Patients who have received prior CAR T cells are eligible. Patients who have received prior BCMA-directed therapy, other than belantamab mafodotin, are eligible. Patients who have received autologous stem cell transplantation >60 days prior are eligible Patients who have received prior allogeneic stem cell transplantation >100 days prior are eligible.
* Female or male patients age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2. PS-3 is permitted if PS is due solely to bone pain.
* Participants must enroll in and comply with the REMS program for pomalidomide.
* Fulfil the criteria for Adequate Organ System Function Based on Safety Assessments

  °Hematologic
* Absolute neutrophil count (ANC)a ≥1.0 × 10^9/L
* Hemoglobin a ≥8.0 g/dL
* Platelets a ≥50 × 10^9/L

  °Hepatic
* Total bilirubin ≤1.5 × ULN; (isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%)
* ALT ≤ 2.5 × ULN °Renal
* eGFRb ≥30 mL/min^b
* Spot urine (albumin/creatinine ratio from spot urine) ≤ 500 mg/g (56 mg/mmol) OR Urine dipstick Negative/trace (if ³1+ only eligible if confirmed <500 mg/g (56 mg/mmol) by albumin/creatinine ratio (spot urine from first void)

  °Cardiac
* Left Ventricular Ejection Fraction (LVEF) by ECHO ≥40% Note: Laboratory results obtained during Screening should be used to determine eligibility criteria. In situations where laboratory results are outside the permitted range, the Investigator may re-test the participant and the subsequent within range screening result may be used to confirm eligibility.

  1. Without Growth factor support for the past 14 days, excluding erythropoietin. Transfusions are allowed
  2. As calculated by the CKD-EPI formula.
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤ 1,with the exception of peripheral neuropathy attributable to bortezomib.
* Female participants: A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

  ° Is not a woman of childbearing potential (WOCBP)
* Nonchildbearing potential is defined as follows (by other than medical reasons):

  ° 45 years of age and has not had menses for >1 year
* Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
* Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.

OR

* Is a WOCBP and agrees to use a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency, during the intervention period and for at least 6 months after the last dose of study intervention.
* WOCBP must have a negative serum or urine pregnancy test within 72 hours prior to treatment with nirogacestat and must agree to use a highly effective method of contraception (i.e. copper-containing intrauterine device, established use of oral, inserted, injected or implanted hormonal method of contraception, or male/female sterilization, etc.)
* WOCBP must agree not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with a nearly undetected pregnancy.

* Male participants: Male participants are eligible to participate if they agree to the following during the intervention period and for 6 months after the last dose of study treatment to allow for clearance of any altered sperm: Male patients must use a condom when having sexual intercourse with a woman of childbearing potential(WOCBP) while receiving treatment with nirogacestat and for at least 6 months after the last dose. An additional form of highly effective contraception should also be used by the female partner, if of child-bearing potential
* Signed and dated Informed Consent by study participant.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other procedures.

Exclusion Criteria:

* Prior treatment with belantamab mafodotin
* Systemic anti-myeloma therapy (including systemic steroids) within ≤14 days, or plasmapheresis within 7 days prior to the first dose of study drug.
* Use of an investigational drug within 14 days or five half-lives (whichever is longer) preceding the first dose of study drug.
* Prior treatment with a monoclonal antibody within 30 days of receiving the first dose of study drugs.
* Radiation therapy within 2 weeks prior to study entry (bone lesions requiring radiation may be treated with limited [i.e., ≤ 25% of bone marrow in field] radiation therapy during this period).
* Patients with a history of stem cell transplant autologous within 60 days or allogeneic within 100 days prior to study enrollment.
* Patients with AL amyloidosis will be excluded.
* Participant must not have had major surgery ≤4 weeks prior to initiating study treatment.
* Evidence of active mucosal or internal bleeding.
* Presence of active renal condition (infection or requirement for dialysis). Participants with isolated proteinuria resulting from multiple myeloma are eligible, provided they fulfill criteria given
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, or otherwise stable chronic liver disease per investigator's assessment).
* Participants with invasive malignancies other than multiple myeloma are excluded, unless the second malignancy has been considered medically stable for at least 2years. The participant must not be receiving active therapy, other than hormonal therapy for this disease with the exceptions of successfully treated non-metastatic basal cell, squamous cell skin carcinoma, or in-situ carcinoma.
* Evidence of cardiovascular risk including any of the following:

  * Evidence of current clinically significant untreated arrhythmias, including clinically significant ECG abnormalities including 2nd degree (Mobitz Type II) or3rd degree atrioventricular (AV) block.
  * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 3 months of Screening
  * Class III or IV heart failure as defined by the New York Heart Association functional classification system.
  * Uncontrolled hypertension
* Known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs chemically related to belantamab mafodotin, or any of the components of the study treatment.
* Pregnant or lactating female.
* Active infection requiring treatment.
* Participant has known human immunodeficiency virus (HIV) infection, unless the participant can meet all of the following criteria:

  1. Established anti-retroviral therapy (ART) for at least 4 weeks and HIV viral load<400 copies/mL, and
  2. CD4+ T-cell (CD4+) counts ≥350 cells/μL, and
  3. No history of acquired immunodeficiency s-defining opportunistic infections within the last 12 months.

Note: Consideration must be given to ART and prophylactic antimicrobials that may have a drug-drug interaction and/or overlapping toxicities with belantamab mafodotin or other combination products as relevant.

* Presence of hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb at Screening or within 3 months prior to first dose of study treatment). Note: Participants with positive Hepatitis B antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis B RNA test is obtained.
* Positive hepatitis C antibody test result or positive hepatitis C RNA test result at Screening or within 3 months prior to first dose of study treatment. Note: Participants with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained. Hepatitis RNA testing is optional and participants with negative Hepatitis C antibody test are not required to also undergo Hepatitis C RNA testing
* Current corneal disease except for mild punctate keratopathy. Note: Participants with mild punctate keratopathy are allowed.
* Participant must not use contact lenses while participating in this study.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
* Study participant has known malabsorption syndrome or preexisting gastrointestinal conditions that may impair absorption of nirogacestat (e.g., gastric bypass, lap band, or other gastric procedures that would alter absorption); delivery of nirogacestat via nasogastric tube or gastrostomy tube is not allowed.
* Concomitant administration of a strong or moderate CYP3A4 inhibitor or inducer within14 days prior to first dose of nirogacestat including foods such as seville oranges, grapefruit or hybrid. Please note that strong or moderate CYP3A inhibitor or inducer administration is to be prohibited during participation on study.
* Concomitant administration of a strong CYP1A2 inhibitors while on treatment with pomalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experienced Dose-Limiting Toxicities (DLTs) | up to six weeks
  The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized.

SECONDARY OUTCOMES:
Clinical Response | 2 years
  Traditional Response Criteria from International Myeloma Working Group Criteria for Multiple Myeloma

CONTACTS AND LOCATIONS:
Overall Officials: Malin Hultcrantz, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to:crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org